CLINICAL TRIAL: NCT04264117
Title: Comparison of Contact-force Monitoring Irrigated Tip Catheter and Mesh-like Irrigated Tip Catheter in Atrial Fibrillation Ablation: Prospective Randomized Trial (COMMIC Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2017-0019
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Atrial Fibrillation ablation; Prospective randomized trial
MeSH Terms: conditions — Atrial Fibrillation | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FlexAbility (Mesh-like irrigated tip catheter) group (Active Comparator)
  Interventions: Procedure: FlexAbility (Mesh-like irrigated tip catheter) group
- TactiCath (Contract force monitoring catheter) group (Experimental)
  Interventions: Procedure: TactiCath (Contract force monitoring catheter) group

INTERVENTIONS:
Procedure: FlexAbility (Mesh-like irrigated tip catheter) group — 1. AF catheter ablation (PV isolation and linear ablations)
  2. 30 sec ablation in each point
  3. 35W in anterior LA, 30 W in posterior LA
  4. Irrigation flow rate 13mL/min
  5. Measuring procedure time, Ablation time
  6. Rhythm follow-up based on guidelines
  Arms: FlexAbility (Mesh-like irrigated tip catheter) group
Procedure: TactiCath (Contract force monitoring catheter) group — 1. AF catheter ablation (PV isolation and linear ablations)
  2. contact force >10g, target force-time integral 400 in each point
  3. 35W in anterior LA, 30 W in posterior LA
  4. Irrigation flow rate 15mL/min at 30W ablation, 30mL/min at 35W ablation
  5. Measuring procedure time, Ablation time
  6. Rhythm follow-up based on guidelines
  Arms: TactiCath (Contract force monitoring catheter) group

SUMMARY:
Mesh-type flexible tip (MFT) catheter is developed to generate bigger radiofrequency (RF) lesion, and contract force (CF) catheter improves the maintenance of catheter-tissue contact during atrial fibrillation catheter ablation (AFCA).

The investigators compared clinical outcome of AFCA conducted by MFT catheter and CF catheter in prospective randomized manner.

The investigators prospectively assigned 230 patients with AF in a 1:1 ratio to ablation by MFT catheter (FlexAbility™, Abbott Inc. USA) and CF catheter (TactiCath™, Abbott Inc. USA). The primary end point was AF recurrence after single procedure, and the secondary end point was response to antiarrhythmic drugs.

DETAILED DESCRIPTION:
A. Study design

1. Prospective randomization (FlexAbility group vs. TactiCath group )
2. Target number of subjects: 360 (180 per group)
3. Rhythm follow-up : 2012 ACC/AHA/ESC guidelines (Holter monitoring at the baseline, 2 month, and thereafter every 6 months; ECG if the patient has any symptom)
4. Anticoagulant therapy followed by 2014 ACC/AHA/ESC guidelines
5. All complications in each group will be evaluated including the re-hospitalization rate, cardioversion frequency, major cardiovascular event, and mortality rate.

B. Progress and rhythm/ECG follow-up

1. To be performed in accordance with the 2012 ACC/AHA/HRS guidelines for AF management
2. Follow-up at 2 weeks, 2 months, and thereafter every 6-month.
3. Rhythm control at 2 months, and thereafter every 6-month follow-up with Holter
4. If the patient complains of symptoms, ECG will be performed at any time, and rhythm follow-up will be carried out with a Holter or event recorder.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate indiction for AF catheter ablation (20~80 years old)
* Echocardiographically measured left atrial size < 55mm
* Anticoagulation eligible patients

Exclusion Criteria:

* AF associated with significant cardiac anomaly, structural heart disease affecting hemodynamics
* Ineligible to CT imaging due to significant renal disease
* Prior history of AF catheter ablation or cardiac surgery
* Active internal bleeding
* Anticoagulation ineligible patients
* Valvular AF
* Life expectancy < 1year
* Drug or alcohol addicted patients
* Other unacceptable patients for clinical trial determined by investigators

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
procedure related complication rate - open heart surgery, stroke, pericardial tamponade, groin complication, and other procedure related complications within a month | 1 month after the procedure
clinical recurrence rate of AF or AT lasting > 30s. Regular rhythm follow-up based on 2012 ACC/AHA/HRS guidelines | 12 months after the procedure
clinical recurrence rate of AF or AT lasting > 30s. Regular rhythm follow-up based on 2012 ACC/AHA/HRS guidelines | 24 months after the procedure
Major cardiovascular events - death, myocardial infarction, coronary angioplasty, stroke, arrhythmia or heart failure related admission | 12 months after the procedure
Major cardiovascular events - death, myocardial infarction, coronary angioplasty, stroke, arrhythmia or heart failure related admission | 24 months after the procedure

SECONDARY OUTCOMES:
procedure time | intraoperative
RF energy delivery time | within 30 minutes after the procedure
volume of irrigated saline infusion | within 30 minutes after the procedure
post-procedural readmission rate | 12 months after the procedure
post-procedural readmission rate | 24 months after the procedure
post-procedural cardioversion rate | 12 months after the procedure
post-procedural cardioversion rate | 24 months after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided